CLINICAL TRIAL: NCT05964608
Title: The Effect of Behavioral Therapy Given to Men With Premature Ejaculation on Symptoms and Their Partners' Sexual Functioning and Sexual Quality of Life
Brief Title: The Effect of Behavioral Therapy Given to Men and Their Partners'
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Ece Kaplan, Asst. Prof., University of Gaziantep
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GAUN-EBE-EK-01
Record Dates: First submitted 2023-07-17; First posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Premature Ejaculation; Sexual Function Disturbances
MeSH Terms: conditions — Premature Ejaculation; Sexual Dysfunctions, Psychological | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Pre-tests were applied to the men (Personal Information Form and PEDT) and their spouses (Personal Information Form, FSFI, and SQOL-F) just before the behavioral treatment was applied to the men in the treatment group. In the first interview with the men, the researchers delivered information about behavioral therapy and set therapy days and hours. Structured interviews, consisting of a total of 6 sessions, were held once every two weeks for men with premature ejaculation problems. Behavioral therapy took place once every two weeks for a total of six 45-minute sessions. The "stop-start technique" was the therapy used. Behavioral therapy interviews were conducted at the urology outpatient clinic of the hospital. Post-tests were administered to men with premature ejaculation (PEDT) and their spouses (FSFI and SQOL-F) immediately after the 6th session was completed.
  Interventions: Behavioral: Behavioral Therapy

INTERVENTIONS:
Behavioral: Behavioral Therapy — Structured interviews, consisting of a total of 6 sessions, were held once every two weeks for men with premature ejaculation problems. Behavioral therapy took place once every two weeks for a total of six 45-minute sessions. The "stop-start technique" was the therapy used. Behavioral therapy interviews were conducted at the urology outpatient clinic of the hospital. Post-tests were administered to men with premature ejaculation (PEDT) and their spouses (FSFI and SQOL-F) immediately after the 6th session was completed.

SUMMARY:
Premature ejaculation involves not only sexual problems but also relationship and communication difficulties, and behavioral approaches to the treatment of premature ejaculation are promising.

DETAILED DESCRIPTION:
Introduction and hypothesis: Premature ejaculation potentially affects not only men but also their partners negatively. The null hypothesis for this study is Behavioral therapy given to men with premature ejaculation has no effect on the symptoms and their partners' sexual functions and quality of sexual life.

Methods: A quasi-experimental study. The current study was conducted in 84 men and their partners. The "Personal Information Form", "Premature Ejaculation Diagnostic Tool (PEDT)", "Female Sexual Function Index (FSFI)", and "Sexual Quality of Life-Female (SQOL-F)" were used to collect data. Behavioral therapy, consisting of a total of 6 sessions of 45 minutes, was applied once every two weeks.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate
* Having no communication barriers
* Literacy
* Age 18-45 years
* Having no diagnosis of sexual dysfunctions
* Having no medical illnesses (psychiatric diseases, pelvic anatomical disorder, post-menopause, etc.) that might affect the sexual function
* Having a spouse diagnosed with premature ejaculation according to DSM-5 criteria
* Having a spouse without any prior behavioral therapy for premature ejaculation
* Being a man diagnosed with lifelong premature ejaculation according to the ISSM criteria.
* Being married

Exclusion Criteria:

-Men and their partners who did not meet all inclusion criteria were excluded from the present study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Premature Ejaculation Diagnostic Tool (PEDT) | six weeks
  it was developed by Symonds et al. (2007) to better define premature ejaculation for use in clinical studies, this is a 5-point Likert-type scale consisting of 5 items. The scale was adapted to Turkish by Serefoglu et al. (2009). The highest score that can be obtained from the scale is 20.0 and the lowest score is 0.0. Scores higher than 11 are defined as "PE", scores of 9-10 are defined as "possible PE", and scores of eight or less are defined as "no PE".

SECONDARY OUTCOMES:
Female Sexual Function Index (FSFI) | six weeks
  Developed by Rosen et al. in 2000, the Female Sexual Function Index (FSFI) is a multidimensional scale consisting of six sections and 19 items evaluating female sexual function. The scale was adapted to Turkish by Aygin and Eti Aslan (2005). The scale contains six sub-dimensions: desire, arousal, lubrication (wetting), orgasm, satisfaction, and pain. The highest score that can be obtained from the scale is 36.0 and the lowest is 2.0. As the score obtained from the scale increases, sexual function improves. The simple mathematical algorithm calculation is organized to determine the scoring of the subscales and the entire scale. Factor loads were determined as 0.6 for desire, 0.3 for arousal and lubrication, and 0.4 for orgasm, satisfaction, and pain.
Sexual Quality of Life-Female (SQOL-F) | six weeks
  It was developed by Symonds et al. in 2005, the Sexual Quality of Life-Female (SQOL-F) is a six-point Likert-type questionnaire consisting of 18 items to evaluate women's sexual quality of life. Tugut and Golbasi (2010) adapted the questionnaire to Turkish in 2010. Each item addresses sexual life over the preceding four weeks. The questionnaire uses a 1-6 point system (1-totally agree, 2-strongly agree, 3-somewhat disagree, 5-strongly disagree, 6-totally disagree), and the range of points that can be obtained is between 18 and 108. As the score obtained from the questionnaire increases, the quality of sexual life increases.

CONTACTS AND LOCATIONS:
Overall Officials: Kazım Doğan, Dr., Principal Investigator — Istinye University
Locations (1):
- ECE, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No